CLINICAL TRIAL: NCT04338737
Title: A Randomized Controlled Study of Early Versus Delayed Oral Post Operative Feeding After Cesarean Section
Brief Title: Post Operative Feeding After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, sarah mohamed hassan, assisstant professor of obstetrcs and gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS-235-2019
Record Dates: First submitted 2020-04-01; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Feeding Patterns
Keywords: early feeding ,late feeding
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fluid and soft food (Active Comparator): It consists of 100 patients that will be allocated for early post-operative oral feeding receiving water and clear fluid approximately 2 hours after surgery, followed by soft food and regular diet 4 hours later irrespective to intestinal sounds, flatus or stool.
  Interventions: Other: timming of feeding
- fluid only (Active Comparator): It consists of 100 patients that will be allocated for early Postoperative oral feeding receiving water and clear fluid approximately 2 hours after surgery till the return of intestinal sounds, then soft food and regular diet later on.
  Interventions: Other: timming of feeding
- Npo (Active Comparator): It consists of 100 patients that will receive no oral feeding till passage of flatus instead 2 to 3 Litres of intravenous fluid will be used for feeding. Water and fluid will be then offered, followed by soft foods and then a regular diet.
  Interventions: Other: timming of feeding

INTERVENTIONS:
Other: timming of feeding — post-operative oral feeding receiving water and clear fluid after surgery, followed by soft food and regular diet

SUMMARY:
3 different post ceseraen secton feeding regmen are compared

DETAILED DESCRIPTION:
300 women admitted to the labor and delivery unit in kasr Elainy teaching hospital, Following the decision to perform a cesarean section because of obstetric indications. The study involved only elective cesarean sections.

The 300 patients participated in this work and will be randomly and equally divided into three groups:

1. Group A :

   It consists of 100 patients that will be allocated for early post-operative oral feeding receiving water and clear fluid approximately 2 hours after surgery, followed by soft food and regular diet 4 hours later irrespective to intestinal sounds, flatus or stool.
2. Group B :

   It consists of 100 patients that will be allocated for early Postoperative oral feeding receiving water and clear fluid approximately 2 hours after surgery till the return of intestinal sounds, then soft food and regular diet later on.
3. Group C :

It consists of 100 patients that will receive no oral feeding till passage of flatus instead 2 to 3 Litres of intravenous fluid will be used for feeding. Water and fluid will be then offered, followed by soft foods and then a regular diet.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age from 20 to 40.
* Primigravida and previous 1 or two cesarean section.
* Elective cesarean section.
* Regional anaesthesia.
* Singleton pregnancy

Exclusion Criteria:

* Medical disorders as (sever preeclampsia, diabetes, liver or kidney diseases).
* Intraoperative intestinal injury.
* Previous major abdominal surgery except cesarean section.
* Obstructed labor with

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
duration minutes till return of bowel sound | time interval in minutes from the end of surgery till the return of intestinal sound
  hearing of intestinal sound
maternal satisfaction from time of initiation of oral feeding after caesarean section. | before discharge from hospital (range of 24 hours)
  Assessment of patient satisfaction before discharge from hospital using visual analogue scale.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP